CLINICAL TRIAL: NCT00123344
Title: Atrial Pacing for Termination and Prevention of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Anne M. Gillis M.D., University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15099
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Bradycardia; Atrial Fibrillation
Keywords: symptomatic bradycardia; paroxysmal atrial fibrillation; antitachycardia pacing therapies; prevention algorithms
MeSH Terms: conditions — Bradycardia; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Device: AT501 pacemaker

SUMMARY:
Atrial fibrillation (AF) is the most common sustained arrhythmia and is associated with substantial morbidity and mortality. Present treatment strategies are aimed at termination of AF and prevention of AF recurrence using antiarrhythmic drugs or heart rate control drugs. Drugs are not always well tolerated, so atrial pacing as a strategy for prevention of atrial tachyarrhythmias is being explored.

The AT501 pacemaker has both "prevention" and "treatment" algorithms for atrial tachyarrhythmias. The investigators wish to determine whether these special features, over the long term, decrease the amount of time the person experiences AF.

DETAILED DESCRIPTION:
There are some clinical and experimental data to suggest that atrial overdrive pacing should prevent AF. In our pacemaker population with tachy-brady syndrome, and in the PA3 study population, we observed that AF frequently clusters and may recur early following an episode of AF.

We are conducting a randomized trial of both prevention algorithms and antitachycardia pacing (ATP) therapies for the treatment of atrial tachyarrhythmias and thereby prevention of AF over the longterm.

Patients with a history of paroxysmal AF who received an AT501 pacemaker for the treatment of bradycardia will be randomized to having both the prevention and therapy algorithms "ON", both "OFF" or having only the therapy algorithms "ON". They will be followed every 3 months for 1 year, then every 6 months for an 2 additional years. Recurrence and frequency of AF will be determined over time based on data retrieved from the device at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Reason for pacing: symptomatic bradycardia
* Paroxysmal AF (>5 min duration, >3 episodes) post implant of AT501 pacemaker
* On stable antiarrhythmic drugs
* Life expectancy >3 years

Exclusion Criteria:

* Life expectancy <3 years
* Unable to give informed consent
* Unable to come for followup
* Chronic AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1999-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To determine the effects of antitachycardia pacing (ATP) therapies on prevention of atrial fibrillation recurrence over the long term

SECONDARY OUTCOMES:
To determine the effects of atrial pacing prevention algorithms on the time to recurrence of atrial fibrillation over the long term

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Gillis, MD, Principal Investigator — University of Calgary, Professor of Medicine; D. George Wyse, MD, Ph.D, Study Chair — University of Calgary, Professor of Medicine; John M Rothschild, MD, Study Chair — University of Calgary, Professor of Medicine; M Sarah Rose, Ph D, Study Chair — University of Calgary, Statistician
Locations (1):
- Foothills Hospital, Calgary, Alberta, Canada